CLINICAL TRIAL: NCT04476043
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study of the Efficacy and Safety of INCB054707 in Participants With Hidradenitis Suppurativa
Brief Title: To Assess the Efficacy and Safety of INCB054707 in Participants With Hidradenitis Suppurativa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INCB 54707-204; 2020-001981-13 (EudraCT Number)
Record Dates: First submitted 2020-07-15; First posted 2020-07-17 (Actual); Results first posted 2023-01-26 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Hidradenitis Suppurativa; Acne Inversa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- INCB054707 15 mg (Experimental): Participants will receive INCB054707 15 milligrams (mg) for 16 weeks in the Placebo-controlled Treatment Period, followed by INCB054707 75 mg for 36 weeks in the Open-label Extension Period. Participants will have the option to continue open-label treatment for an additional 48 weeks.
  Interventions: Drug: INCB054707
- INCB054707 45 mg (Experimental): Participants will receive INCB054707 45 mg for 16 weeks in the Placebo-controlled Treatment Period, followed by INCB054707 75 mg for 36 weeks in the Open-label Extension Period. Participants will have the option to continue open-label treatment for an additional 48 weeks.
  Interventions: Drug: INCB054707
- INCB054707 75 mg (Experimental): Participants will receive INCB054707 75 mg for 52 weeks in the Placebo-controlled Treatment Period (16 weeks) plus the Open-label Extension Period (36 weeks). Participants will have the option to continue open-label treatment for an additional 48 weeks.
  Interventions: Drug: INCB054707
- Placebo followed by INCB054707 75 mg (Placebo Comparator): Participants will receive placebo for 16 weeks in the Placebo-controlled Treatment Period, followed by INCB054707 75 mg for 36 weeks in the Open-label Extension Period. Participants will have the option to continue open-label treatment for an additional 48 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: INCB054707 — Oral; Tablet
  Other Names: Povorcitinib
  Arms: INCB054707 15 mg; INCB054707 45 mg; INCB054707 75 mg
Drug: Placebo — Oral; Tablet
  Arms: Placebo followed by INCB054707 75 mg

SUMMARY:
To evaluate the efficacy and safety of INCB054707 in participants with hidradenitis suppurativa over a 16-week placebo-controlled treatment period followed by a 36-week open-label extension period. All eligible participants will be invited to continue treatment for an additional 48-week Long-term extension period (also open label).

ELIGIBILITY:
Inclusion Criteria:

* HS disease duration of at least 3 months before screening.
* Willingness to avoid pregnancy or fathering children.
* Active HS in at least 2 distinct anatomical areas.
* Participants agree NOT to use topical antiseptics on the areas affected by HS lesions during the placebo-controlled 16-week treatment period

Exclusion Criteria:

* Draining fistula count of > 20 at screening or baseline.
* Women who are pregnant (or who are considering pregnancy) or lactating.
* Medical history including thrombocytopenia, coagulopathy or platelet dysfunction, Q-wave interval abnormalities, current or history of certain infections, cancer, lymphoproliferative disorders and other medical conditions at the discretion of the investigator.
* History of failure to treatment of inflammatory diseases with JAK inhibitors.
* Have evidence of active or latent or inadequately treated infection with Mycobacterium tuberculosis.
* Participants known to be infected with HIV, Hepatitis B, or Hepatitis C.
* Laboratory values outside of the protocol-defined ranges.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2023-08-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (40):
- United States (25):
  - Investigative Site 005, Hoover, Alabama
  - Investigative Site 003, Gilbert, Arizona
  - Investigative Site 011, Phoenix, Arizona
  - Investigative Site 014, Fountain Valley, California
  - Investigative Site 010, Fremont, California
  - Investigative Site 012, Huntington Beach, California
  - Investigative Site 022, Newbury Park, California
  - Investigative Site 009, Sacramento, California
  - Investigative Site 025, Cromwell, Connecticut
  - Investigative Site 015, Coral Gables, Florida
  - Investigative Site 021, Miami, Florida
  - Investigative Site 006, Tampa, Florida
  - Investigative Site 001, Tampa, Florida
  - Investigative Site 016, Atlanta, Georgia
  - Investigative Site 002, West Lafayette, Indiana
  - Investigative Site 027, Baton Rouge, Louisiana
  - Investigative Site 023, New Orleans, Louisiana
  - Investigative Site 013, Boston, Massachusetts
  - Investigative Site 004, Fort Gratiot, Michigan
  - Investigative Site 019, St Louis, Missouri
  - Investigative Site 026, The Bronx, New York
  - Investigative Site 008, Chapel Hill, North Carolina
  - Investigative Site 017, Winston-Salem, North Carolina
  - Investigative Site 007, Hershey, Pennsylvania
  - Investigative Site 018, Bellaire, Texas
- Canada (2):
  - Investigative Site 101, Calgary, Alberta
  - Investigative Site 102, Calgary, Alberta
- Investigative Site 304, Nantes, France
- Germany (6):
  - Investigative Site 403, Berlin
  - Investigative Site 401, Bochum
  - Investigative Site 405, Dessau
  - Investigative Site 406, Dresden
  - Investigative Site 404, Erlangen
  - Investigative Site 402, Frankfurt am Main
- Poland (3):
  - Investigative Site 552, Rzeszów
  - Investigative Site 551, Wroclaw
  - Investigative Site 553, Wroclaw
- Spain (3):
  - Investigative Site 703, Granada
  - Investigative Site 702, Madrid
  - Investigative Site 701, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 209 participants were enrolled at 36 study centers: 26 in North America and 10 in Europe. Data are reported through the cut-off date of 15 December 2021.
Groups:
- Placebo: Participants received oral placebo once a day (QD) for 16 weeks in the Placebo-controlled Treatment Period.
- INCB054707 15 mg: Participants received oral INCB054707 15 milligrams (mg) QD for 16 weeks in the Placebo-controlled Treatment Period.
- INCB054707 45 mg: Participants received oral INCB054707 45 mg QD for 16 weeks in the Placebo-controlled Treatment Period.
- INCB054707 75 mg: Participants received oral INCB054707 75 mg QD for 16 weeks in the Placebo-controlled Treatment Period.
Period: Overall Study
Arm/Group | Placebo | INCB054707 15 mg | INCB054707 45 mg | INCB054707 75 mg
Started | 52 | 52 | 52 | 53
Completed | 48 | 47 | 45 | 51
Not Completed | 4 | 5 | 7 | 2
Not completed — Withdrawal by Subject | 1 | 3 | 4 | 1
Not completed — Lost to Follow-up | 1 | 1 | 2 | 1
Not completed — Adverse Event | 2 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | INCB054707 15 mg | INCB054707 45 mg | INCB054707 75 mg | Total
Number analyzed (Participants) | 52 | 52 | 52 | 53 | 209
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (9.96) | 38.2 (10.85) | 37.3 (12.51) | 37.5 (10.83) | 37.1 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 37 | 39 | 39 | 158
  Male | 9 | 15 | 13 | 14 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 40 | 36 | 35 | 36 | 147
  Black/African American | 10 | 13 | 12 | 16 | 51
  Asian | 1 | 2 | 2 | 1 | 6
  American Indian/Alaska Native | 0 | 0 | 1 | 0 | 1
  Captured as Other | 1 | 1 | 2 | 0 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 5 | 7 | 6 | 28
  Not Hispanic or Latino | 41 | 47 | 44 | 47 | 179
  Unknown | 1 | 0 | 0 | 0 | 1
  Captured as Other | 0 | 0 | 1 | 0 | 1
Mean abscess and inflammatory nodule (AN) count [Mean (Standard Deviation); unit: abscesses and inflammatory nodules] | 11.2 (5.85) | 11.8 (7.10) | 12.9 (12.34) | 10.6 (7.24) | 11.6 (8.48)
Mean International Hidradenitis Suppurativa Severity Score System (IHS4) score [Mean (Standard Deviation); unit: scores on a scale] — The IHS4 is a composite, dynamic score and validated tool used to determine Hidradenitis Suppurativa severity. It employs a weighted scale using the number of inflammatory nodules, the number of abscesses, and the number of draining tunnels (fistulas or sinuses), with respective weight factors of 1, 2, and 4. Scores: mild=0-3; moderate=4-10; severe ≥11.
  scores on a scale | 22.9 (17.02) | 22.4 (23.24) | 23.5 (22.79) | 18.9 (17.25) | 21.9 (20.21)
Mean abscess, inflammatory nodule (IN), and draining fistula (DF) (ANF) count [Mean (Standard Deviation); unit: abscesses, INs, and DFs] | 13.6 (6.36) | 14.1 (10.08) | 15.1 (13.51) | 12.2 (8.94) | 13.7 (10.03)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Abscess and Inflammatory Nodule (AN) Count at Week 16
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The mixed model repeated measure (MMRM) included the fixed effects of treatment group (placebo and INCB054707 15, 45, and 75 mg), stratification factors (disease severity [Hurley Stage I, II, and III] and geographical region [North America and outside of North America]), visit (Weeks 2, 4, 6, 8, 12, and 16), treatment by visit interaction, and covariates of Baseline measurement and Baseline measurement by visit interaction. The variance-covariance matrix of the within-participant errors in MMRM are modeled as unstructured.
Time Frame: Baseline; Week 16
Population: Intent-to-Treat (ITT) Population: all randomized participants. Treatment groups for this population were defined according to the treatment assignment at randomization. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: abscesses and inflammatory nodules
Arm/Group | Placebo | INCB054707 15 mg | INCB054707 45 mg | INCB054707 75 mg
Number analyzed (Participants) | 43 | 45 | 43 | 46
abscesses and inflammatory nodules | -2.5 (0.88) | -5.2 (0.86) | -6.9 (0.88) | -6.3 (0.85)
Statistical Analysis 1: Comparison: Placebo vs INCB054707 15 mg; Test type: Superiority; p = 0.0277, MMRM; Least squares mean (LSM) difference = -2.7, 95% CI 2-sided [-5.2 to -0.3], Standard Error of Mean 1.23
Statistical Analysis 2: Comparison: Placebo vs INCB054707 45 mg; Test type: Superiority; p = 0.0006, MMRM; LSM difference = -4.4, 95% CI 2-sided [-6.8 to -1.9], Standard Error of Mean 1.25
Statistical Analysis 3: Comparison: Placebo vs INCB054707 75 mg; Test type: Superiority; p = 0.0021, MMRM; LSM difference = -3.8, 95% CI 2-sided [-6.2 to -1.4], Standard Error of Mean 1.22

2. Secondary Outcome: Percentage of Participants Who Achieved a Hidradenitis Suppurativa Clinical Response (HiSCR) at Week 16
Description: HiSCR, the key secondary endpoint, was defined as at least a 50% decrease from Baseline in AN count with no increase in the number of abscesses or draining fistulas.
Time Frame: Baseline; Week 16
Population: ITT Population. 95% confidence interval (CI) was based on the Clopper-Pearson exact method. Missing post-Baseline values were imputed as nonresponders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | INCB054707 15 mg | INCB054707 45 mg | INCB054707 75 mg
Number analyzed (Participants) | 52 | 52 | 52 | 53
percentage of participants | 28.8 [17.1 to 43.1] | 48.1 [34.0 to 62.4] | 44.2 [30.5 to 58.7] | 45.3 [31.6 to 59.6]
Statistical Analysis 1: Comparison: Placebo vs INCB054707 15 mg; Test type: Superiority; p = 0.0445, Wald test; Odds Ratio (OR) = 2.3, 95% CI 2-sided [1.0 to 5.3] — Logistic regression model with treatment group and stratification factors (disease severity and geographical region)
Statistical Analysis 2: Comparison: Placebo vs INCB054707 15 mg; Test type: Superiority; Difference in response rate = 19.2, Standard Error of Mean 9.35 — Standard error of difference between response rates was from normal approximation
Statistical Analysis 3: Comparison: Placebo vs INCB054707 45 mg; Test type: Superiority; p = 0.0998, Wald test; Odds Ratio (OR) = 2.0, 95% CI 2-sided [0.9 to 4.6] — Logistic regression model with treatment group and stratification factors (disease severity and geographical region)
Statistical Analysis 4: Comparison: Placebo vs INCB054707 45 mg; Test type: Superiority; Difference in response rate = 15.4, Standard Error of Mean 9.32 — Standard error of difference between response rates was from normal approximation
Statistical Analysis 5: Comparison: Placebo vs INCB054707 75 mg; Test type: Superiority; p = 0.0829, Wald test; Odds Ratio (OR) = 2.1, 95% CI 2-sided [0.9 to 4.7] — Logistic regression model with treatment group and stratification factors (disease severity and geographical region)
Statistical Analysis 6: Comparison: Placebo vs INCB054707 75 mg; Test type: Superiority; Difference in response rate = 16.4, Standard Error of Mean 9.29 — Standard error of difference between response rates was from normal approximation

3. Secondary Outcome: Percentage of Participants Who Achieved a HiSCR at Weeks 2 Through 12
Description: HiSCR was defined as at least a 50% decrease from Baseline in AN count with no increase in the number of abscesses or draining fistulas.
Time Frame: Baseline; Weeks 2, 4, 6, 8, and 12
Population: ITT Population. 95% CI was based on the Clopper-Pearson exact method. Missing post-Baseline values were imputed as nonresponders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | INCB054707 15 mg | INCB054707 45 mg | INCB054707 75 mg
Number analyzed (Participants) | 52 | 52 | 52 | 53
percentage of participants
  Week 2 | 15.4 [6.9 to 28.1] | 25.0 [14.0 to 38.9] | 34.6 [22.0 to 49.1] | 34.0 [21.5 to 48.3]
  Week 4 | 25.0 [14.0 to 38.9] | 36.5 [23.6 to 51.0] | 44.2 [30.5 to 58.7] | 49.1 [35.1 to 63.2]
  Week 6 | 17.3 [8.2 to 30.3] | 32.7 [20.3 to 47.1] | 48.1 [34.0 to 62.4] | 52.8 [38.6 to 66.7]
  Week 8 | 28.8 [17.1 to 43.1] | 36.5 [23.6 to 51.0] | 44.2 [30.5 to 58.7] | 52.8 [38.6 to 66.7]
  Week 12 | 30.8 [18.7 to 45.1] | 42.3 [28.7 to 56.8] | 48.1 [34.0 to 62.4] | 58.5 [44.1 to 71.9]

4. Secondary Outcome: Percentage of Participants Who Achieved HiSCR75 From Weeks 2 to 16
Description: HiSCR75 was defined as at least a 75% decrease from Baseline in AN count with no increase in the number of abscesses or draining fistulas.
Time Frame: Baseline; Weeks 2, 4, 6, 8, 12, and 16
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | INCB054707 15 mg | INCB054707 45 mg | INCB054707 75 mg
Number analyzed (Participants) | 52 | 52 | 52 | 53
percentage of participants
  Week 2 | 1.9 [0.0 to 10.3] | 9.6 [3.2 to 21.0] | 13.5 [5.6 to 25.8] | 18.9 [9.4 to 32.0]
  Week 4 | 7.7 [2.1 to 18.5] | 15.4 [6.9 to 28.1] | 21.2 [11.1 to 34.7] | 15.1 [6.7 to 27.6]
  Week 6 | 9.6 [3.2 to 21.0] | 17.3 [8.2 to 30.3] | 28.8 [17.1 to 43.1] | 24.5 [13.8 to 38.3]
  Week 8 | 19.2 [9.6 to 32.5] | 23.1 [12.5 to 36.8] | 30.8 [18.7 to 45.1] | 35.8 [23.1 to 50.2]
  Week 12 | 19.2 [9.6 to 32.5] | 26.9 [15.6 to 41.0] | 32.7 [20.3 to 47.1] | 39.6 [26.5 to 54.0]
  Week 16 | 17.3 [8.2 to 30.3] | 30.8 [18.7 to 45.1] | 28.8 [17.1 to 43.1] | 30.2 [18.3 to 44.3]

5. Secondary Outcome: Mean Change From Baseline in the Severity of the Disease, as Assessed by the International Hidradenitis Suppurativa Severity Score System (IHS4) Score, From Weeks 2 to 16
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The IHS4 is a composite, dynamic score and validated tool used to determine Hidradenitis Suppurativa severity. It employs a weighted scale using the number of inflammatory nodules, the number of abscesses, and the number of draining tunnels (fistulas or sinuses), with respective weight factors of 1, 2, and 4. Scores: mild=0-3; moderate=4-10; severe ≥11. MMRM included the fixed effects of treatment group (placebo and INCB054707 15, 45, and 75 mg), stratification factors (disease severity [Hurley Stage I, II, and III] and geographical region [North America and outside of North America]), visit (Weeks 2, 4, 6, 8, 12, and 16), treatment by visit interaction, and covariates of Baseline measurement and Baseline measurement by visit interaction. The variance-covariance matrix of the within-participant errors in MMRM are modeled as unstructured.
Time Frame: Baseline; Weeks 2, 4, 6, 8, 12, and 16
Population: ITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | INCB054707 15 mg | INCB054707 45 mg | INCB054707 75 mg
Number analyzed (Participants) | 52 | 52 | 52 | 53
scores on a scale
  Week 2: number analyzed (Participants) | 47 | 51 | 48 | 52
  Week 2 | -2.4 (1.17) | -3.8 (1.13) | -6.7 (1.16) | -6.1 (1.12)
  Week 4: number analyzed (Participants) | 49 | 50 | 50 | 52
  Week 4 | -2.1 (1.52) | -3.9 (1.49) | -9.3 (1.51) | -9.3 (1.47)
  Week 6: number analyzed (Participants) | 45 | 47 | 48 | 49
  Week 6 | -3.1 (1.77) | -4.7 (1.73) | -10.7 (1.75) | -10.6 (1.71)
  Week 8: number analyzed (Participants) | 45 | 50 | 47 | 51
  Week 8 | -3.0 (1.85) | -4.0 (1.79) | -11.8 (1.83) | -10.7 (1.78)
  Week 12: number analyzed (Participants) | 45 | 45 | 45 | 49
  Week 12 | -3.1 (1.80) | -5.5 (1.76) | -11.8 (1.79) | -11.9 (1.73)
  Week 16: number analyzed (Participants) | 43 | 45 | 43 | 46
  Week 16 | -3.1 (1.96) | -5.6 (1.92) | -11.0 (1.96) | -12.1 (1.90)

6. Secondary Outcome: Percentage of Participants Who Achieved AN50, AN75, AN90, and AN100 From Weeks 2 to 16
Description: AN50, AN75, AN90, and AN100 were defined as at least a 50%, 75%, 90%, and 100% decrease, respectively, from Baseline in AN count.
Time Frame: Baseline; Weeks 2, 4, 6, 8, 12, and 16
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | INCB054707 15 mg | INCB054707 45 mg | INCB054707 75 mg
Number analyzed (Participants) | 52 | 52 | 52 | 53
percentage of participants
  AN50, Week 2 | 15.4 [6.9 to 28.1] | 25.0 [14.0 to 38.9] | 34.6 [22.0 to 49.1] | 39.6 [26.5 to 54.0]
  AN50, Week 4 | 30.8 [18.7 to 45.1] | 44.2 [30.5 to 58.7] | 46.2 [32.2 to 60.5] | 58.5 [44.1 to 71.9]
  AN50, Week 6 | 32.7 [20.3 to 47.1] | 46.2 [32.2 to 60.5] | 51.9 [37.6 to 66.0] | 56.6 [42.3 to 70.2]
  AN50, Week 8 | 36.5 [23.6 to 51.0] | 55.8 [41.3 to 69.5] | 53.8 [39.5 to 67.8] | 54.7 [40.4 to 68.4]
  AN50, Week 12 | 44.2 [30.5 to 58.7] | 51.9 [37.6 to 66.0] | 55.8 [41.3 to 69.5] | 62.3 [47.9 to 75.2]
  AN50, Week 16 | 36.5 [23.6 to 51.0] | 55.8 [41.3 to 69.5] | 57.7 [43.2 to 71.3] | 52.8 [38.6 to 66.7]
  AN75, Week 2 | 1.9 [0.0 to 10.3] | 9.6 [3.2 to 21.0] | 13.5 [5.6 to 25.8] | 20.8 [10.8 to 34.1]
  AN75, Week 4 | 7.7 [2.1 to 18.5] | 15.4 [6.9 to 28.1] | 23.1 [12.5 to 36.8] | 18.9 [9.4 to 32.0]
  AN75, Week 6 | 13.5 [5.6 to 25.8] | 25.0 [14.0 to 38.9] | 32.7 [20.3 to 47.1] | 26.4 [15.3 to 40.3]
  AN75, Week 8 | 21.2 [11.1 to 34.7] | 28.8 [17.1 to 43.1] | 32.7 [20.3 to 47.1] | 37.7 [24.8 to 52.1]
  AN75, Week 12 | 23.1 [12.5 to 36.8] | 32.7 [20.3 to 47.1] | 36.5 [23.6 to 51.0] | 39.6 [26.5 to 54.0]
  AN75, Week 16 | 17.3 [8.2 to 30.3] | 36.5 [23.6 to 51.0] | 36.5 [23.6 to 51.0] | 34.0 [21.5 to 48.3]
  AN90, Week 2 | 0.0 [0.0 to 6.8] | 3.8 [0.5 to 13.2] | 1.9 [0.0 to 10.3] | 11.3 [4.3 to 23.0]
  AN90, Week 4 | 0.0 [0.0 to 6.8] | 5.8 [1.2 to 15.9] | 7.7 [2.1 to 18.5] | 5.7 [1.2 to 15.7]
  AN90, Week 6 | 5.8 [1.2 to 15.9] | 5.8 [1.2 to 15.9] | 11.5 [4.4 to 23.4] | 9.4 [3.1 to 20.7]
  AN90, Week 8 | 5.8 [1.2 to 15.9] | 15.4 [6.9 to 28.1] | 19.2 [9.6 to 32.5] | 18.9 [9.4 to 32.0]
  AN90, Week 12 | 5.8 [1.2 to 15.9] | 17.3 [8.2 to 30.3] | 13.5 [5.6 to 25.8] | 20.8 [10.8 to 34.1]
  AN90, Week 16 | 3.8 [0.5 to 13.2] | 17.3 [8.2 to 30.3] | 19.2 [9.6 to 32.5] | 18.9 [9.4 to 32.0]
  AN100, Week 2 | 0.0 [0.0 to 6.8] | 3.8 [0.5 to 13.2] | 1.9 [0.0 to 10.3] | 7.5 [2.1 to 18.2]
  AN100, Week 4 | 0.0 [0.0 to 6.8] | 3.8 [0.5 to 13.2] | 5.8 [1.2 to 15.9] | 5.7 [1.2 to 15.7]
  AN100, Week 6 | 0.0 [0.0 to 6.8] | 3.8 [0.5 to 13.2] | 7.7 [2.1 to 18.5] | 9.4 [3.1 to 20.7]
  AN100, Week 8 | 3.8 [0.5 to 13.2] | 13.5 [5.6 to 25.8] | 11.5 [4.4 to 23.4] | 17.0 [8.1 to 29.8]
  AN100, Week 12 | 3.8 [0.5 to 13.2] | 13.5 [5.6 to 25.8] | 11.5 [4.4 to 23.4] | 18.9 [9.4 to 32.0]
  AN100, Week 16 | 3.8 [0.5 to 13.2] | 15.4 [6.9 to 28.1] | 11.5 [4.4 to 23.4] | 17.0 [8.1 to 29.8]

7. Secondary Outcome: Mean Change From Baseline in AN Count at Weeks 2 to 12
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value. MMRM included the fixed effects of treatment group (placebo and INCB054707 15, 45, and 75 mg), stratification factors (disease severity [Hurley Stage I, II, and III] and geographical region [North America and outside of North America]), visit (Weeks 2, 4, 6, 8, 12, and 16), treatment by visit interaction, and covariates of Baseline measurement and Baseline measurement by visit interaction. The variance-covariance matrix of the within-participant errors in MMRM are modeled as unstructured.
Time Frame: Baseline; Weeks 2, 4, 6, 8, and 12
Population: ITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: abscesses and inflammatory nodules
Arm/Group | Placebo | INCB054707 15 mg | INCB054707 45 mg | INCB054707 75 mg
Number analyzed (Participants) | 52 | 52 | 52 | 53
abscesses and inflammatory nodules
  Week 2: number analyzed (Participants) | 47 | 51 | 48 | 52
  Week 2 | -1.7 (0.69) | -2.7 (0.66) | -3.4 (0.69) | -4.0 (0.66)
  Week 4: number analyzed (Participants) | 49 | 50 | 50 | 52
  Week 4 | -3.0 (0.71) | -3.6 (0.70) | -4.8 (0.71) | -5.3 (0.69)
  Week 6: number analyzed (Participants) | 45 | 47 | 48 | 49
  Week 6 | -2.7 (0.77) | -4.8 (0.76) | -5.3 (0.77) | -6.2 (0.75)
  Week 8: number analyzed (Participants) | 45 | 50 | 47 | 51
  Week 8 | -2.7 (0.82) | -4.7 (0.79) | -6.4 (0.82) | -5.7 (0.79)
  Week 12: number analyzed (Participants) | 45 | 45 | 45 | 49
  Week 12 | -2.8 (0.84) | -5.0 (0.82) | -6.7 (0.84) | -6.5 (0.81)

8. Secondary Outcome: Percentage of Participants With a Total AN Count of 0 to 2 From Weeks 2 to 16
Description: Total AN count was assessed throughout the study.
Time Frame: Weeks 2, 4, 6, 8, 12, and 16
Population: ITT Population. Only participants with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | INCB054707 15 mg | INCB054707 45 mg | INCB054707 75 mg
Number analyzed (Participants) | 52 | 52 | 52 | 53
percentage of participants
  Week 2: number analyzed (Participants) | 47 | 51 | 48 | 52
  Week 2 | 4.3 | 9.8 | 16.7 | 23.1
  Week 4: number analyzed (Participants) | 49 | 50 | 50 | 52
  Week 4 | 14.3 | 20.0 | 20.0 | 23.1
  Week 6: number analyzed (Participants) | 45 | 47 | 48 | 49
  Week 6 | 13.3 | 19.1 | 31.3 | 38.8
  Week 8: number analyzed (Participants) | 45 | 50 | 47 | 51
  Week 8 | 28.9 | 30.0 | 38.3 | 41.2
  Week 12: number analyzed (Participants) | 45 | 45 | 45 | 49
  Week 12 | 28.9 | 33.3 | 46.7 | 38.8
  Week 16: number analyzed (Participants) | 43 | 45 | 43 | 46
  Week 16 | 25.6 | 44.4 | 51.2 | 37.0

9. Secondary Outcome: Mean Change From Baseline in Draining Fistula Count From Weeks 2 to 16
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Weeks 2, 4, 6, 8, 12, and 16
Population: ITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: draining fistulas
Arm/Group | Placebo | INCB054707 15 mg | INCB054707 45 mg | INCB054707 75 mg
Number analyzed (Participants) | 52 | 52 | 52 | 53
draining fistulas
  Baseline | 2.4 (3.97) | 2.3 (4.44) | 2.2 (4.04) | 1.6 (2.85)
  Change from Baseline at Week 2: number analyzed (Participants) | 47 | 51 | 48 | 52
  Change from Baseline at Week 2 | -0.2 (1.23) | -0.2 (1.01) | -0.6 (1.62) | -0.2 (1.30)
  Change from Baseline at Week 4: number analyzed (Participants) | 49 | 50 | 50 | 52
  Change from Baseline at Week 4 | 0.0 (1.80) | 0.0 (1.11) | -0.8 (2.59) | -0.6 (2.44)
  Change from Baseline at Week 6: number analyzed (Participants) | 45 | 47 | 48 | 49
  Change from Baseline at Week 6 | -0.2 (2.14) | 0.1 (1.85) | -1.0 (2.95) | -0.8 (2.62)
  Change from Baseline at Week 8: number analyzed (Participants) | 45 | 50 | 47 | 51
  Change from Baseline at Week 8 | -0.2 (2.46) | 0.2 (2.10) | -1.1 (2.82) | -0.8 (2.70)
  Change from Baseline at Week 12: number analyzed (Participants) | 45 | 45 | 45 | 49
  Change from Baseline at Week 12 | -0.3 (2.17) | 0.0 (2.71) | -1.0 (2.87) | -1.0 (2.61)
  Change from Baseline at Week 16: number analyzed (Participants) | 43 | 45 | 43 | 46
  Change from Baseline at Week 16 | -0.3 (2.05) | 0.1 (3.25) | -0.8 (3.20) | -1.1 (2.57)

10. Secondary Outcome: Mean Change From Baseline in Abscess, Inflammatory Nodule (IN), and Draining Fistula (DF) (ANF) Count From Weeks 2 to 16
Description: as for outcome 7
Time Frame: Baseline; Weeks 2, 4, 6, 8, 12, and 16
Population: ITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: abscesses, INs, and DFs
Arm/Group | Placebo | INCB054707 15 mg | INCB054707 45 mg | INCB054707 75 mg
Number analyzed (Participants) | 52 | 52 | 52 | 53
abscesses, INs, and DFs
  Week 2: number analyzed (Participants) | 47 | 51 | 48 | 52
  Week 2 | -1.8 (0.74) | -2.9 (0.72) | -4.0 (0.74) | -4.4 (0.71)
  Week 4: number analyzed (Participants) | 49 | 50 | 50 | 52
  Week 4 | -2.7 (0.83) | -3.5 (0.82) | -5.7 (0.82) | -6.2 (0.80)
  Week 6: number analyzed (Participants) | 45 | 47 | 48 | 49
  Week 6 | -2.6 (0.92) | -4.7 (0.90) | -6.4 (0.92) | -7.1 (0.89)
  Week 8: number analyzed (Participants) | 45 | 50 | 47 | 51
  Week 8 | -2.6 (0.96) | -4.4 (0.93) | -7.5 (0.96) | -6.8 (0.92)
  Week 12: number analyzed (Participants) | 45 | 45 | 45 | 49
  Week 12 | -2.7 (0.99) | -5.0 (0.97) | -7.7 (0.98) | -7.6 (0.95)
  Week 16: number analyzed (Participants) | 43 | 45 | 43 | 46
  Week 16 | -2.4 (1.06) | -5.1 (1.03) | -7.7 (1.05) | -7.6 (1.02)

11. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. An AE could have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. A TEAE was defined as any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug until the end of the safety follow-up.
Time Frame: up to Week 16
Population: Safety Population: all participants who received at least 1 dose of INCB054707 or placebo during the Placebo-controlled Period
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | INCB054707 15 mg | INCB054707 45 mg | INCB054707 75 mg
Number analyzed (Participants) | 52 | 52 | 50 | 53
Participants | 34 | 31 | 30 | 32

ADVERSE EVENTS:
Time Frame: up to Week 16
Description: Treatment-emergent adverse events (TEAEs), defined as AEs either reported for the first time or the worsening of pre-existing events after the first dose of study drug until the end of the safety follow-up, have been reported for members of the Safety Population (all participants who received at least 1 dose of INCB054707 or placebo during the Placebo-controlled Period).
Arm/Group | Placebo | INCB054707 15 mg | INCB054707 45 mg | INCB054707 75 mg
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52 | 0/50 | 0/53
Serious Adverse Events (participants affected / at risk) | 3/52 | 2/52 | 1/50 | 0/53
Other Adverse Events (participants affected / at risk) | 15/52 | 20/52 | 17/50 | 19/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=52) | INCB054707 15 mg (N=52) | INCB054707 45 mg (N=50) | INCB054707 75 mg (N=53)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=52) | INCB054707 15 mg (N=52) | INCB054707 45 mg (N=50) | INCB054707 75 mg (N=53)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (5) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) | 3 (3)
Fatigue (General disorders) | 4 (4) | 5 (5) | 6 (6) | 6 (6)
Headache (Nervous system disorders) | 5 (5) | 4 (5) | 3 (3) | 4 (4)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (6) | 3 (3) | 2 (2) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 4 (4)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/43/NCT04476043/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/43/NCT04476043/SAP_001.pdf